CLINICAL TRIAL: NCT02006771
Title: A Randomized Crossover Trial to Compare the Changes of Postprandial Oxidative Stress After Consumption of Meals From Different Cultures in Healthy Chinese Adults
Brief Title: Cultural Meal and Postprandial Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ruth Chan, Research assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 461813; 461813 (Other Grant/Funding Number: GRF)
Record Dates: First submitted 2013-11-28; First posted 2013-12-10 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Oxidative Stress
Keywords: Meal; Postprandial oxidative stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Southern Chinese meal (Experimental): White rice (1 bowl), stir fried Choi sum (0.5 bowl) and stir fried lean pork (0.5 bowl) cooked with maize oil
  Interventions: Other: Southern Chinese meal
- Northern Chinese meal (Experimental): Noodles (1 bowl) and shredded pork with sweet bean sauce (0.5 bowl) cooked with blend oil
  Interventions: Other: Northern Chinese meal
- American meal (Experimental): Hamburger with cheese (1 piece), French fries (117 g) cooked with canola blend oil plus Coca-cola classic (21 fluid ounces)
  Interventions: Other: American meal
- South Indian meal (Experimental): Basmati rice (1 bowl), chicken curry dish (0.5 bowl), dry vegetable dish (i.e. green beans mixed with herbs) (0.5 bowl), yogurt made with milk powder mainly (0.5 bowl), pickle made with lemon, salt, chilli powder, Asafoetida and vegetable based oil (1 tablespoon)
  Interventions: Other: South Indian meal

INTERVENTIONS:
Other: Southern Chinese meal — White rice (1 bowl), stir fried choi sum (0.5 bowl) and stir fried lean pork (0.5 bowl) cooked with maize oil
  Arms: Southern Chinese meal
Other: Northern Chinese meal — Noodles (1 bowl) and shredded pork with sweet bean sauce (0.5 bowl) cooked with blend oil
  Arms: Northern Chinese meal
Other: American meal — Hamburger with cheese (1 piece), French fries (117 g) cooked with canola blend oil and Coca-cola classic (21 fluid ounces)
  Arms: American meal
Other: South Indian meal — Basmati rice (1 bowl), chicken curry dish (0.5 bowl), dry vegetable dish (i.e. green beans mixed with herbs) (0.5 bowl), yogurt made with milk powder mainly (0.5 bowl), pickle made with lemon, salt, chilli powder, Asafoetida and vegetable based oil (1 tablespoon)
  Arms: South Indian meal

SUMMARY:
This one-year randomized crossover study is proposed to compare the changes of postprandial oxidative stress (POS) after consumption of meals from different cultures in healthy Chinese adults, using a 'real-life, cultural meal' approach. It is hypothesized that the changes of POS differ with meals from different cultures. Four cultural meals are chosen, namely Southern Chinese, Northern Chinese, American, and South Indian, based on the known prevalence of chronic diseases between Caucasians, Chinese and Indians, and within the Southern and Northern Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy male or female of Chinese ethnicity with BMI less than 25 kg/m2
* Aged from 18 to 45 years for female to avoid menopausal effect, and 18 to 50 years for male (inclusive)
* Normal glucose tolerance as assessed by fasting HbA1c of <6% at the screening
* Willing to give consent and follow the study procedures

Exclusion Criteria:

* Lifestyle factors that affect POS as shown by the literature including
* Current smoker
* Physically active as defined by three days or more of 30 minutes [accumulated over the course of a day] moderate to vigorous activity weekly in the past three months. Vigorous physical activity is described as causing heavy sweating or a large increase in breathing or heart rate, and moderate as causing light sweating or a slight to moderate increase in breathing or heart rate.
* Regular or current use of vitamin or antioxidant supplements
* Pregnant or lactating
* Concurrent participation in any clinical trial or dietary intervention program
* Adherence to a special diet, allergies or aversions to foods on the study meals
* Use of medications that could affect study outcomes
* With diabetes, hypertension, renal, liver or thyroid dysfunction, any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of plasma allantoin from 0 (pre-meal) to 6 hours post-meal | pre-meal (0 hour), 2, 4, 6 hours post-meal

SECONDARY OUTCOMES:
Change of urine F2-isoprostanes from 0 (pre-meal) to 6 hours post-meal | pre-meal (0 hour), 2, 4, 6 hours post-meal

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Chan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China